CLINICAL TRIAL: NCT06660160
Title: Evaluating The Feasibility And Safety Of A Group Exercise Program Supported By Audiovisual Media During Hemodialysis (GrExID)
Brief Title: Group Exercise Program Supported By Audiovisual Media During Hemodialysis
Acronym: GrExID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: B.Braun Avitum AG (Industry); Universidade Federal de Juiz de Fora (Unknown)
Responsible Party: Principal Investigator, Eva Segura Ortí, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrExID
Record Dates: First submitted 2024-10-18; First posted 2024-10-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Failure; Hemodialysis; Sarcopenia; Functional Capacity; Muscle Strength Dynamometer; Physical Activity Level
Keywords: Chronic Kidney Failure; Hemodialysis; Exercise; Sarcopenia; Muscle strength; Functional capacity; Dynamometer; Physical activity level
MeSH Terms: conditions — Kidney Failure, Chronic; Sarcopenia; Motor Activity | interventions — Exercise; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): Patients over 18 years old of both sexes, who have been undergoing HD for at least three months, generally in three sessions per week that are in the room that was randomized to do exercise.
  Interventions: Other: Exercise program supported by audiovisual media
- Control Group (CG) (No Intervention): Patients over 18 years old of both sexes, who have been undergoing HD for at least three months, generally in three sessions per week that are in the room that was randomized to will continue with the usual treatment.

INTERVENTIONS:
Other: Exercise program supported by audiovisual media — The intervention group will perform the group exercise protocol during HD sessions. The videos with the exercises will be broadcast on all televisions simultaneously, so that the volunteers perform the exercises along with the person in the video.
  * The first level of difficulty includes 5 exercises for the lower limbs and 3 exercises for the upper limbs. One set of 10 repetitions will be performed for each exercise per session.
  * The second level includes 3 exercises for the lower limbs and 2 exercises for the upper limbs. These consist of proprioceptive neuromuscular facilitation diagonals for both the lower and upper limbs. One set of 10 repetitions will be performed for each exercise, once per week, for 3 weeks.
  * The third level includes 8 combined lower and upper limb exercises performed simultaneously. One set of 20 repetitions will be performed for each exercise.
  Exercises will be performed 3 times per week over a 4-week period, for a total of 12 planned exercise sessions.
  Other Names: Exercise; Exercise training; Exercise training during hemodialysis; Physiotherapy; Online exercise training
  Arms: Intervention Group (IG)

SUMMARY:
People with chronic kidney disease (CKD) undergoing hemodialysis (HD) experience muscular complications, such as sarcopenia, which worsen their functional capacity and increase mortality. Exercise programs during HD are an effective strategy to combat sedentary behavior, and implementing them through innovative technologies could facilitate their adoption in clinics, benefiting more patients. Therefore, the study's objectives are to assess the feasibility and safety of a group exercise program supported by audiovisual media conducted during HD sessions. Additionally, it will analyze factors influencing adherence, identify potential causes for interruptions or failure to perform the prescribed exercise, and evaluate the risk and prevalence of sarcopenia, its association with low muscle strength, poor muscle quality, and physical inactivity.

DETAILED DESCRIPTION:
A 4-week randomized experimental study will be conducted, using an exercise protocol during HD, broadcast simultaneously on television. The frequency of exercise completion, reasons for non-completion, adverse events, as well as sarcopenia, muscle strength, muscle characteristics through ultrasound and electrical bioimpedance, and physical activity levels will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old of both sexes;
* Undergoing HD for at least three months in three sessions per week, four hours, totaling 12 hours per week.

Exclusion Criteria:

* Lower limb amputations;
* Neurological, musculoskeletal, or osteoarticular disorders;
* Severe and unstable comorbidities;
* Undergoing high doses of corticosteroids (>30 mg/day);
* Inability to understand the measurement methods used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Safety Assessment | From start to finish of intervention (4 weeks)
  Feasibility will be assessed through adherence rate (number of sessiones performed out of sessions offered).
Feasibility and Safety Assessment | From start to finish of intervention (4 weeks)
  Adverse events of the exercise during the study (number of adverse events)

SECONDARY OUTCOMES:
Sarcopenia Risk Assessment | It will be applied before and after the 4 weeks of intervention.
  The risk of sarcopenia will be evaluated using the SARC-F (Strength, Assistance with walking, Rising from a chair, Climbing stairs and Falls )questionnaire. Score ranges from 0 a 10, higher scores mean higher risc of sarcopenia.
Muscle Strength Assessment | It will be applied before and after the 4 weeks of intervention
  Handgrip strength
Muscle Strength Assessment | It will be applied before and after the 4 weeks of intervention.
  Lower limb muscle strength assessments via digital manual dynamometry will be performed during HD using the MMT Lafayette Instrument Company hand dynamometer.
Muscle Characteristics | It will be applied before and after the 4 weeks of intervention
  The quantity and quality of muscle mass will be evaluated by the cross-sectional area of the rectus femoris muscle, measured by muscle ultrasound.
Muscle Characteristics | It will be applied before and after the 4 weeks of intervention.
  Body composition and appendicular skeletal muscle mass will also be measured by multi-frequency bioelectrical impedance analysis (BIA),
Physical Activity Level Assessment | It will be applied before and after the 4 weeks of intervention.
  The level of physical activity will be evaluated using the HAP questionnaire (Average Activity Score AAS).

CONTACTS AND LOCATIONS:
Locations (1):
- B. Braun Avitum - Centro de Atención Renal, Massamagrell, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segura-Orti E, Garcia-Testal A. Intradialytic virtual reality exercise: Increasing physical activity through technology. Semin Dial. 2019 Jul;32(4):331-335. doi: 10.1111/sdi.12788. Epub 2019 Mar 27. PMID 30916415
- [Background] Reboredo MM, Neder JA, Pinheiro BV, Henrique DM, Faria RS, Paula RB. Constant work-rate test to assess the effects of intradialytic aerobic training in mildly impaired patients with end-stage renal disease: a randomized controlled trial. Arch Phys Med Rehabil. 2011 Dec;92(12):2018-24. doi: 10.1016/j.apmr.2011.07.190. PMID 22133251
- [Background] Sharma D, Hawkins M, Abramowitz MK. Association of sarcopenia with eGFR and misclassification of obesity in adults with CKD in the United States. Clin J Am Soc Nephrol. 2014 Dec 5;9(12):2079-88. doi: 10.2215/CJN.02140214. Epub 2014 Nov 12. PMID 25392147